CLINICAL TRIAL: NCT00467129
Title: The Role of Genetic Factors in Clinical Outcome for Colorectal Cancer
Brief Title: Genes That Affect Disease Outcome in Patients With Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000540670; SHEFF-SSREC01/271; SHEFF-USMS-SSREC01/271; EU-20727
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Microarray Analysis; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and help doctors understand how patients respond to treatment.

PURPOSE: This clinical trial is examining genes that affect disease outcome in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect blood samples for DNA extraction for genetic studies from patients receiving chemotherapy for metastatic colorectal cancer.
* Collect detailed clinical, pathological, and chemotherapy data from these patients.
* Identify genetic factors that relate to treatment response and outcome in these patients.

OUTLINE: Blood samples are collected and relevant genes and regions are amplified by PCR. PCR products are then sequenced or genotyped for known biological markers and single nucleotide polymorphisms. Tumor samples from surplus pathology specimens are analyzed for expression of candidate genes and mutation in the candidate genes.

Clinical and family history data is also collected by questionnaire.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal cancer
* Currently receiving chemotherapy at Weston Park Hospital

PATIENT CHARACTERISTICS:

* Not Specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2002-07

PRIMARY OUTCOMES:
Survival
Progressive disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Angela Cox, PhD, Study Chair — University of Sheffield